CLINICAL TRIAL: NCT00901303
Title: Pilot Study of Abbreviated Chemotherapy Based on Positron Emission Tomography in Hodgkin Lymphoma
Brief Title: Pilot Study of Abbreviated Chemotherapy Based on Positron Emission Tomography (PET) Scan in Hodgkin's Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to lack of accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0810010015
Record Dates: First submitted 2009-04-30; First posted 2009-05-13 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Stage Disease (Other): Group A
  Interventions: Drug: ABVD chemotherapy
- Advance Stage Disease (Other): Group B
  Interventions: Drug: ABVD chemotherapy

INTERVENTIONS:
Drug: ABVD chemotherapy — Adriamycin 25 mg/m2 bleomycin 10 units/m2 vinblastine 6 mg/m2 dacarbazine 375 mg/m on Days 1 and 15 of each 28 day cycle

SUMMARY:
The primary objective of the study is to determine the progression-free survival [PFS] at 36 months for patients with Hodgkin lymphoma who achieve a complete metabolic response as demonstrated by a negative fluorodeoxyglucose (FDG)-PET scan after one cycle of ABVD (adriamycin, bleomycin, vinblastine, dacarbazine) who undergo abbreviated ABVD chemotherapy (3 cycles).

DETAILED DESCRIPTION:
The proposed study is based on the repeated demonstration that patients with Hodgkin lymphoma who attain a negative PET scan early in therapy (after one or 2 cycles of chemotherapy) have a uniformly excellent outcome, with long term disease free survival of 90-95%. We propose to abbreviate chemotherapy in those patients showing a complete metabolic response as measured by FDG-PET after one cycle of ABVD. These patients will undergo two more cycles of ABVD chemotherapy, for a total of 3 cycles. Those patients failing to achieve a complete metabolic response as demonstrated by residual FDG avidity will go off study and be treated as per their primary treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented classical Hodgkin lymphoma according to the WHO Classification. Nodular lymphocyte predominant Hodgkin lymphoma is excluded
* No prior treatment (chemotherapy or radiation therapy) for Hodgkin lymphoma
* Measurable disease must be present either on physical examination or imaging studies. Any tumor mass measurable in two dimensions and > 2 cm is acceptable (or 1.5 cm if 0.5 cm slices are used as in spiral CT scans)
* Age ≥ 18
* Patients must have at least one hypermetabolic lesion identifiable on initial PET scan
* LVEF by ECHO or MUGA within institutional normal limits
* Initial laboratory data should be compatible with the administration of standard doses of ABVD chemotherapy

Exclusion Criteria:

* Patient has no known HIV infection
* Patient is non-pregnant and non-lactating. Due to the teratogenic potential of the agents used in this study, pregnant or nursing women may not be enrolled. Women and men of reproductive potential should agree to use an effective means of birth control
* No other history of lymphoproliferative disorder or granulomatous disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2011-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Elstrom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced Stage Disease: Group B
  ABVD chemotherapy: Adriamycin 25 mg/m2 bleomycin 10 units/m2 vinblastine 6 mg/m2 dacarbazine 375 mg/m on Days 1 and 15 of each 28 day cycle
Period: Overall Study
Arm/Group | Early Stage Disease | Advanced Stage Disease
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Stage Disease | Advanced Stage Disease | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: 36-Month Progression-free Survival Rate
Description: Progression-free survival is defined as the length of time from study intervention to disease progression or death
Time Frame: 36 months
Population: Data was not collected due to early termination of the study.
Groups:
- Group A: early stage disease
  ABVD chemotherapy: Adriamycin 25 mg/m2 bleomycin 10 units/m2 vinblastine 6 mg/m2 dacarbazine 375 mg/m on Days 1 and 15 of each 28 day cycle
- Group B: advanced stage disease
  ABVD chemotherapy: Adriamycin 25 mg/m2 bleomycin 10 units/m2 vinblastine 6 mg/m2 dacarbazine 375 mg/m on Days 1 and 15 of each 28 day cycle
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Zero subjects at risk for adverse events as this was not evaluated due to early study termination.
Arm/Group | Early Stage Disease | Advanced Stage Disease
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No